CLINICAL TRIAL: NCT04029948
Title: Laser Versus Electrical Transurethral Enbloc Resection of Non-muscle Invasive Bladder Tumours: A Randomized Trial
Brief Title: Laser vs. Electorsurgical Enbloc Resection of Bladder Tumours
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmed Elshal, Clinical Professor, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MS.19.07.740
Record Dates: First submitted 2019-07-17; First posted 2019-07-23 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Urinary Bladder Neoplasm
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laser ERBT (Active Comparator): Laser En Bloc Resection Of bladder Tumor
  Interventions: Procedure: Laser En Bloc Resection Of bladder Tumor
- electro-surgical ERBT (Active Comparator): electro-surgical En Bloc Resection Of bladder Tumor
  Interventions: Procedure: Electro-surgical En Bloc Resection Of bladder Tumor

INTERVENTIONS:
Procedure: Laser En Bloc Resection Of bladder Tumor — Using laser beam starting the procedure with circumferential incision few millimetres around the tumour then lifting the tumour and dissection underneath its muscle base
  Arms: laser ERBT
Procedure: Electro-surgical En Bloc Resection Of bladder Tumor — Using electro-surgical loop starting the procedure with circumferential incision few millimetres around the tumour then lifting the tumour and dissection underneath its muscle base
  Arms: electro-surgical ERBT

SUMMARY:
To compare use of electrosurgical energy in doing En Bloc resection of bladder tumours against Laser Energy for En Bloc resection of bladder tumours Patients with non muscle invasive bladder cancer will be enrolled and randomized into either of the two techniques

DETAILED DESCRIPTION:
INTRODUCTION

TURBT [transurethral resection of bladder tumor] constitutes a crucial procedure in the diagnosis and treatment of bladder cancer. A complete resection should be achieved either in fractions in bigger, or en-bloc in smaller tumours. The incise and scattering technique is against all oncological principles, damage caused by heat and fragmentation of the tumour hampers histological processing. The technique of resection in fractions ignores the parameter of negative surgical margins, theoretically, liberating tumour cells into the irrigation fluid, which facilitates their implantation and early recurrence. Furthermore, pathological staging may be impaired.

The absence of lamina muscularis propria (LMP, detrusor muscle, DM) in the specimen is associated with a higher risk of residual disease and early recurrence. Absence of LMP is also associated with lower surgical experience. The frequency of detecting MIBC in the second resection in initial pT1 ranges from 4 to 25%, and increases to 45% when no LMP was present. European guidelines 2018, stated that, En-bloc resection using monopolar or bipolar current, Thulium-YAG or Holmium-YAG laser is feasible in selected exophytic tumours. It provides high quality resected specimens with the presence of detrusor muscle in 96-100% of cases.

Recently, Martin-Doyle et al in the large analysis of 15,215 patients to assess recurrence, progression, and cancer-specific survival (CSS) from 73 studies, the highest impact risk factor was depth of invasion (T1b/c) into lamina propria (progression: [HR], 3.34; P < .001; cancer-specific survival: HR, 2.02; P = .001). Other previously proposed factors also predicted progression and CSS (lymphovascular invasion (LVI), associated CIS, non-use of bacillus Calmette-Guérin (BCG), tumor size > 3 cm, and older age; HRs for progression between 1.32 and 2.88, P ≤ .002; HRs for CSS between 1.28 and 2.08, P ≤ .02).

2018 EUA guidelines stated that, the depth and extent of invasion into the lamina propria (T1 substaging) has been demonstrated to be of prognostic value in retrospective cohort studies (LE: 3). Its use is recommended by the most recent 2016 World Health Organization (WHO) classification. However, the optimal system to substage T1 remains to be defined (Babjuk et al., 2018). These difficulty may be attributed to muscularis mucosa is only identified in 15% to 80% of bladder biopsy specimens, though its presence in 90% of radical cystectomy specimens (Wood, 2012). We have hypothesis that enbloc resection can get muscularis mucosa rate similar to radical cystectomy specimens rate.

In the last decade, the en-bloc resection of bladder tumor (ERBT) as an alternative to TURBT has gained more and more interest among urologists. Theoretically, ERBT offers three goals: to improve the resection quality, lowering perioperative complication rates, and decreasing recurrence rates. A new envisaged goal is also to decrease the number of second TURBTs. By using the correct ERBT technique, higher DM rates in comparison with TURBT can be achieved (theoretically up to 100%)(Kramer et al., 2017) In a recent study with more than 2000 patients of pT1 high-grade tumor, the most important parameter that was associated with recurrence-free survival was the detection of DM within the tissue. The authors stated that in case that DM is present one may even avoid second resections in high-risk NMIBC.

In a retrospective multicentre study (EBRUC) with 221 patients in 4 arms, median tumour size was 2.1 cm and largest tumours reached even 5 cm, with LMP being present in 97.3 %. All techniques have in common that first a circular incision is made in the mucosa around the tumour. Subsequently, the tumour is dissected en-bloc including muscle layer using monopolar/bipolar current or holmium/thulium laser energy. Up to date, no clear answer can be given which patient is suitable for enbloc resection. Roughly, 30% of patients are not eligible because of tumor size, formation, and localization. The challenge of large specimen retrieval could be solved using the combination of vaporisation of the exophytic tumour part and En bloc resection of the tumour ground.

Although bipolar current hypothetically be favorable with regard to the obturator nerve reflex and subsequent bladder perforation (0.9% vs. 6.4%) when compared with monopolar current. In a systematic review and meta-analysis, Cui et al found no statistically significant differences in obturator nerve reflex between bipolar and monopolar TURBT (OR= 0.35; 95% CI, 0.06-1.95; P = 0.23) and also no differences on bladder perforation (OR= 0.51; 95% CI, 0.25-1.01; P = .05). European guidelines 2018, stated that though bipolar resection has been introduced to reduce the risk of complications (e.g., bladder perforation due to obturator nerve stimulation) and to produce better specimens for the pathologist. Currently, the results remain controversial.

Apart from a multitude of retrospective cohort or comparison studies, only two prospective, randomized trials on ERBT have been published. Both studies were performed in China, and details on statistical preparation, patient selection, and definitions of primary and secondary goals are missing. Thus, there is still an urgent need a thoroughly planned trial.

AIMS OF THE WORK

Evaluate the feasibility, safety and efficacy of laser and electrical enbloc resection of non muscle invasive bladder cancer.

Detect exact criteria of tumours eligible for enbloc resection either by laser or electro-surgical energy.

Patients & Methods

I. Study Design:

The design of the research will be a prospective randomised controlled study.

II. Study Setting/Location:

The study will be conducted in a single tertiary centre at Urology and Nephrology Center in Mansoura, Egypt.

Eligible patient presented with visual criteria suggesting NMIBC by outpatient cystoscopy. Patients will be asked to participate in this study and will be provided with an informed consent form in line with Good Clinical Practise and the Declaration of Helsinki.

Recruitment of participants Patients appointed for an outpatient diagnostic cystoscopy will be reviewed for the inclusion and exclusion criteria. Legible patients will be asked to participate in the study and to sign the informed consent form.

Randomisation Randomization will be performed using computer generated random tables using stratified blocked randomization in 1:1 ratio.

peri procedure work up Preoperative evaluations included: detailed medical history, physical examination, routine blood examination, urinalysis & urine cytology, renal and liver function tests, ultrasonography, thoracic radiography, computed tomography with contrast scans of the abdomen and pelvis or MRU, Every patient will undergo cystoscopy.

Intervention All the surgeries will be performed in lithotomy position under spinal or general anesthesia.

One group will be managed by 2-micron wave length laser ERBT while the other group will be managed by electro-surgical ERBT.

Principles of enbloc resection will be applied similarly in both groups by starting the procedure with circumferential incision few millimetres around the tumour then lifting the tumour and dissection underneath its muscle base

VIII. Reporting

1. Surgical reporting

   1. Examination under anesthesia
   2. Pre-resection cytology
   3. Tumor criteria: Site (mapping) , Size (in cm) , Number & Shape
   4. Surgeon perspective about grade of the tumor
   5. Suspected mucosa (CIS)
   6. Resection Data:

   one cut/multiple cuts. Biopsy from the base? Surgeon perspective about resection completion/muscle inclusion or not. Weight of resected tissue.
2. Pathological reporting

   1. Location of the evaluated sample (information obtained from the urologist order form)
   2. Grade of each lesion (by the two systems 1973&2004)
   3. Depth of tumor invasion (T stage)
   4. Presence of concurrent CIS
   5. Presence of detrusor muscle in the specimen
   6. Presence of lymphovascular invasion (LVI)
   7. Presence of unusual histology

IX. Outcome measures:

Primary outcome The primary endpoint for this study is to assess the need of conversion to conventional TURBT Secondary outcomes

Quality of tissue submitted for histopathology assessed by cautery artefact defined as:

Grade 1: Cautery artifacts involving less than one-third of the entire specimen.

Grade 2: Tissue chips with one-third to two-thirds cautery artifacts Grade 3: Tissue chips with over two-thirds cautery artifacts

Peri procedure complications Obturator reflex Bladder perforation as defined by the need of auxiliary drainage procedure or catheter prolongation whenever deemed indicated by the operator Postoperative haematuria, decrease of blood Hb, need for blood transfusion and length of postoperative bladder irrigation Systematic assessment of early postoperative complication by assessing as length of postoperative catheterization and length of hospitalization Recurrence free survival at 1 year. Presence or absence of residual tumours in 2nd look TURBT

STATISTICAL CONSIDERATIONS AND DATA ANALYSIS Sample size and statistical power Based on previous study (Kramer et al., 2015) in which, there was a switch to conventional TURBT in the electrical ERBT group vs laser ERBT (26.3 vs. 1.5 %, respectively), using G*power programme (Universität Düsseldorf) with alpha error 0.05 and power 0.80, total sample size was 100 patients.

Statistical Analysis Continuous data will be summarized using the mean ± SD and compared by t test. Categorical variables will be compared using the χ2 test or Fisher's exact test. The Statistical Package for Social Sciences, version 13.0, for Windows (SPSS, Chicago, IL) will be applied for statistical analysis. P≤.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

Patients presented with visual criteria suggesting NMIBC by outpatient cystoscopy will be legible for inclusion

Exclusion Criteria:

1. Tumor criteria

   1. MIBC
   2. Tumours deemed not legible for Enbloc resection as Judged by the surgeon e.g.

      * location: Tumour in diverticulum, at the anterior wall or close to ureteric orifice….etc
      * Wide base tumour
2. Patients criteria

   1. Bleeding tendency
   2. Synchronous either urethral tumours or upper urinary tract tumours
   3. History of CIS
   4. Contracted bladder

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
number of failed En Bloc resection procedures (need for conversion to conventional resection) | intraoperative
  to assess the need of conversion to conventional Transurethral resection of bladder tumor

SECONDARY OUTCOMES:
number of cases with esidual tumours | 4 weeks postoperative
  Presence or absence of residual tumours during second look bladder biopsy
recurrence rate | 1 year post operative
  rate of tumour recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Elshal, MD, Principal Investigator — Mansoura University
Locations (1):
- Urology and Nprhology Center, Al Mansurah, Aldakahlia, Egypt